CLINICAL TRIAL: NCT01344564
Title: Initiation of Androgen Deprivation Therapy for the Treatment of Prostate Cancer Using Degarelix Acetate Followed by Leuprolide Acetate
Brief Title: Initiation of Androgen Deprivation Therapy for Prostate Cancer Using Degarelix Followed by Leuprolide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Urology of Virginia (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UVA002
Record Dates: First submitted 2011-04-27; First posted 2011-04-29 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Hormone therapy; Testosterone measures
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Leuprolide; luprolide acetate gel depot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ADT (Other): All subjects receive ADT, degarelix acetate for 3 months followed by one 3 month leuprolide depot.
  Interventions: Drug: Degarelix acetate, Leuprolide acetate

INTERVENTIONS:
Drug: Degarelix acetate, Leuprolide acetate — Degarelix acetate, 1 mo depot for 3 months Leuprolide acetate, 3 mo depot once
  Other Names: Firmagon; Eligard

SUMMARY:
The purpose of this study is to determine if patients initiating androgen deprivation therapy (ADT) for prostate cancer can be transitioned from degarelix acetate to leuprolide acetate after an initial three-month period without a rise in serum testosterone. The investigators expect testosterone will quickly and reliably reach castrate levels after initiation of ADT and will remain castrate during the transition, and there will be no "testosterone surge" after leuprolide injection.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Histologically confirmed adenocarcinoma of the prostate
* Androgen deprivation therapy is indicated

Exclusion Criteria:

* Baseline screening serum testosterone <150ng/dL
* Eastern Cooperative Oncology Group (ECOG) score > 2
* Diagnosed spinal or brain metastases
* Hormonal manipulation within previous 6 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Testosterone measurement | 11 times over 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Given, MD, Principal Investigator — Urology of Virginia
Locations (1):
- Urology of Virginia, Virginia Beach, Virginia, United States